CLINICAL TRIAL: NCT03599817
Title: Healthy Lifestyle Promotion Program as a Strategy to Improve Obesity Parameters, Cardiovascular and Metabolic Risk Factors in Yaquis Indigenous in the State of Sonora
Brief Title: Program of Healthy Lifestyle Promotion in Yaqui Indigenous in Sonora
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centro de Investigación en Alimentación y Desarrollo A.C. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: JER002
Record Dates: First submitted 2018-07-16; First posted 2018-07-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2020-01

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy lifestyle promotion program (Experimental): All the participants of the intervention program will be offered group sessions focused on healthy eating, promotion of physical activity and behavioral changes. In this way, the loss of body weight and the increase of physical activity will be promoted. Translating into an improvement in obesity parameters and cardiovascular and metabolic risk factors, to reduce the risk of developing type 2 diabetes.
  Interventions: Behavioral: Healthy lifestyle promotion program

INTERVENTIONS:
Behavioral: Healthy lifestyle promotion program — Before implementing the healthy lifestyle program, it will be adapted according to the characteristics of the Yaqui community, their type of food and the activities they carry out, so that the intervention program is culturally accepted by the community. The intervention will consist of two stages, an intensive phase and a maintenance phase. In the intensive phase, 16 weekly group sessions will be given with the aim of achieving a 5% body weight loss and ensuring that the participants do at least 150 minutes of physical activity per week. In the maintenance phase, 6 monthly group sessions will be given in order to maintain the results achieved in the first stage. In the same maintenance phase, but from 12 to 18 months, the lifestyle trainers will make home visits to the participants. Lifestile trainers will record body weight, physical activity and food consumption. In this period there will be no sessions, only monthly visits.

SUMMARY:
Obesity has become an epidemic worldwide and is considered one of the main causes related to type 2 diabetes. The World Health Organization reported that in 2016, 39% of adults were overweight, while the percentage of obesity was 13%, together 1900 million people were overweight/obese. While in 2014 it was reported that 8.5% of the population in the world suffered from type 2 diabetes. On the other hand, in the national context, the last report of 2016 that 72.5% of the Mexican population suffers from overweight/obesity. In addition, in 2006, 14.4% of Mexicans suffered from type 2 diabetes.

Obesity is a complex chronic state that is developed by an imbalance between the energy ingested and the energy expended. In addition, obesity is considered a chronic inflammatory state of low degree of cause of the immune response generated, as a consequence of the increase of adipose tissue; what explains the imbalance in the markers of inflammation. This inflammation condition has been related to the generation of insulin resistance, the increase in glucose levels and the appearance of various pathologies such as type 2 diabetes and other risk factors for cardiovascular diseases.

The Yaqui ethnic group is located in the center-south zone of the state of Sonora, distributed in 8 traditional villages. A recent study conducted in the Yaqui community reported a prevalence of overweight and obesity of 25% and 43% respectively. In 2008, a prevalence of type 2 diabetes of 18.3% was reported in its inhabitants.

On the other hand, there are successful programs in reducing body weight through interventions aimed at modifying lifestyles such as eating habits and physical function called Lifestyle Modification Programs. These programs have been supported through controlled and randomized clinical trials. Such is the case of the Diabetes Prevention Program. Which has achieved weight reduction and increased physical activity in the subjects treated. The Diabetes Prevention Program has been recognized and adapted for the Centers for Disease Control and Prevention and has been dubbed the "National Diabetes Prevention Program".

The present study is a translational research clinical trial to evaluate the effectiveness of a program to promote the parameters of obesity and diabetes in the cardiovascular communities in the Yaqui community of the state of Sonora.

DETAILED DESCRIPTION:
The study focuses on knowing if the program of promotion of healthy lifestyle can reduce the risk of developing type 2 diabetes in adults of the Yaqui ethnic group with overweight / obesity and with risk of diabetes of the state of Sonora, through the loss of body weight and the promotion of physical activity, in this way to improve obesity parameters and cardiovascular and metabolic risk factors.

The primary hypothesis is that the implementation of a program promoting the healthy lifestyle aimed at adults of the Yaqui ethnic group of Sonora with a diagnosis of overweight or obesity and a Finnish Diabetes Risk Score (FINDRISC) ≥12 will significantly improve in the medium term (12 months) the body weight, triglycerides, fasting glucose and interleukin-6 (IL-6).

The secondary hypotheses will be as follows: the implementation of a program to promote a healthy lifestyle aimed at adults of the Yaqui ethnic group of Sonora with a diagnosis of overweight or obesity, and FINDRISC score ≥12 will improve significantly in the short term (6 months) obesity parameters, blood glucose levels, insulin, lipid profile, blood pressure and physical activity.

The implementation of a healthy lifestyle promotion program aimed at adults of the Sonoran Yaqui ethnic group with a diagnosis of overweight or obesity and a FINDRISC score ≥12 will significantly improve medium-term (12 months) obesity parameters, blood levels of insulin, lipid profile, inflammation markers, blood pressure and physical activity.

The implementation of a healthy lifestyle promotion program aimed at adults of the Sonoran Yaqui ethnic group with a diagnosis of overweight or obesity and a FINDRISC score ≥12 will significantly improve long-term (18 months) obesity parameters, blood levels, lipid profile, blood pressure and physical activity.

.

ELIGIBILITY:
Inclusion Criteria:

* Men and women being of the Yaqui tribe
* Age 20 years and less than 65
* Overweight or obese (BMI ≥25 kg/m2)
* FINDRISC score of 12 or higher
* Sign up the consent form and wish to participate

Exclusion Criteria:

* Subjects with diagnosis previous of diabetes
* Uncontrolled hypertension (systolic blood pressure ≥160 mmHg and diastolic blood pressure ≥100 mmHg)
* Renal insufficiency
* Hepatopathies
* Neoplasms
* Inflammatory and traumatic rheumatoid arthritis
* Cardiovascular disease
* Chronic obstructive pulmonary disease
* Thyroid disease
* Systemic lupus erythematosus
* Inflammatory bowel disease
* HIV
* Psoriasis
* Mesangial proliferative glomerulonephritis
* Seriously ill
* Bacterial and viral infections at the time of taking the blood sample
* Pregnant women and/or stage of lactation
* Subjects with limitations to carry out physical exercise
* Subjects that have participated in another similar program
* Subjects in pharmacological treatment for obesity
* People under pharmacological treatment that alter glucose tolerance and lipid levels

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-07-24 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Body weight (kg) | Change in body weight from baseline to 6 months and change in body weight from baseline to 12 months
  Change in body weight
Triglycerides (mg/dL) | Change in triglycerides from baseline to 6 months and change in triglycerides baseline to 12 months
  Change in triglycerides
Fasting glucose (mg/dL) | Change in fasting glucose from baseline to 6 months and change in fasting glucose from baseline to 12 months
  Change in fasting glucose
IL-6 (pg/ml) | Change in IL-6 from baseline to 12 months
  Change in IL-6

SECONDARY OUTCOMES:
Body Mass Index (kg/m2) | Change in Body Mass Index from baseline to 6 months and change in Body Mass Index from baseline to 12 months
  Change in Body Mass Index
Waist circumference (cm) | Change in waist circumference from baseline to 6 months and change in waist circumference from baseline to 12 months
  Change in waist circumference
Body fat percentage (%) | Change in body fat percentage from baseline to 6 months and change in body fat percentage from baseline to 12 months
  Change in body fat percentage
Fasting insulin (mg/dL) | Change in fasting insulin from baseline to 6 months and change in fasting insulin from baseline to 12 months
  Change in fasting insulin
Total cholesterol (mg/dL) | Change in total cholesterol from baseline to 6 months and change in total cholesterol from baseline to 12 months
  Change in total cholesterol
LDL-cholesterol (mg/dL) | Change in LDL-cholesterol from baseline to 6 months and change in LDL-cholesterol from baseline to 12 months
  Change in LDL-cholesterol
HDL-cholesterol (mg/dL) | Change in HDL-cholesterol from baseline to 6 months and change in HDL-cholesterol from baseline to 12 months
  Change in HDL-cholesterol
Systolic and diastolic blood pressure (mmHg) | Change in systolic and diastolic blood pressure from baseline to 6 months and change in systolic and diastolic blood pressure from baseline to 12 months
  Change in systolic and diastolic blood pressure
Physical activity (minutes/week) | Change in physical activity from baseline to 6 months and change in physical activity from baseline to 12 months
  Change in physical activity
Tumor Necrosis Factor-α (TNF-α) (pg/ml) | Change in TNF-α from baseline to 12 months
  Change in TNF-α
Adiponectin (µg/ml) | Change in adiponectin from baseline to 12 months
  Change in adiponectin
Body weight (kg) | Change in body weight from 6 months to 12 and 18 months
  Change in body weight
Body Mass Index (kg/m2) | Change in body mass index from 6 months to 12 and 18 months
  Change in body mass index
Waist circumference (cm) | Change in waist circumference from 6 months to 12 and 18 months
  Change in waist circumference
Body fat percentage (%) | Change in waist circumference from 6 months to 12 and 18 months
  Change in body fat percentage
Fasting glucose (mg/dL) | Change in fasting glucose from 6 months to 12 and 18 months
  Change in fasting glucose
Total cholesterol (mg/dL) | Change in total cholesterol from 6 months to 12 and 18 months
  Change in total cholesterol
LDL-cholesterol (mg/dL) | Change in LDL-cholesterol from 6 months to 12 and 18 months
  Change in LDL-cholesterol
HDL-cholesterol (mg/dL) | Change in HDL-cholesterol from 6 months to 12 and 18 months
  Change in HDL-cholesterol
Systolic and diastolic blood pressure (mmHg) | Change in systolic and diastolic blood pressure from 6 months to 12 and 18 months
  Change in systolic and diastolic blood pressure
Physical activity (minutes/week) | Change in physical activity from 6 months to 12 and 18 months
  Change in physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Julián Esparza-Romero, Ph.D, Principal Investigator — Centro de Investigación en Alimentación y Desarrollo
Locations (4):
- Mexico (4):
  - Dispensario médico, Ciudad Obregón, Loma de Guamúchil
  - Dispensario médico, Guaymas, Pótam
  - Dispensario médico, Guaymas, Tórim
  - Dispensario médico, Guaymas, Vícam

IPD SHARING:
Plan to Share IPD: Undecided